CLINICAL TRIAL: NCT01483443
Title: Prophylactic Oophorectomy Followed by Chemotherapy Versus Chemotherapy Alone in Colorectal Patients With or Without Ovarian Metastasis
Brief Title: Oophorectomy Followed by Chemotherapy Versus Chemotherapy Alone in Colorectal Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Won-Suk Lee, Assistant Prof, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIRBA2263
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Stage IV Colon Cancer
Keywords: oophrectomy; survival
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oophrectomy group (Experimental): Patient undergone oophrectomy along with primary tumor
  Interventions: Procedure: Oophrectomy
- without oophrectomy (No Intervention): Patient group without oophrectomy

INTERVENTIONS:
Procedure: Oophrectomy — Both oophrectomy
  Other Names: No other intervention needed
  Arms: Oophrectomy group

SUMMARY:
This is a prospective phase III trial to define the role of oophorectomy in metastatic colorectal cancer patients with ovarian metastasis.

DETAILED DESCRIPTION:
A recent study demonstrated that colorectal cancer with ovarian metastases were less responsive to chemotherapy compared to extraovarian metastases. The survival impact of oophorectomy has not been defined yet in this clinical setting. The incidence of microscopic ovarian metastasis has been reported to be approximately 10%. Therefore, the investigators propose a prospective study of oophorectomy followed by standard chemotherapy versus standard chemotherapy alone to determine whether oophorectomy increases survival.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18
2. histologically confirmed adenocarcinoma of colon
3. documented ovarian metastasis in CT or MRI or PET-CT
4. advanced (stage IV), metastatic, or recurrent
5. ECOG performance status of 0~2
6. adequate marrow, hepatic, renal and cardiac functions
7. no prior surgical treatment to ovary
8. provision of a signed written informed consent

Exclusion Criteria:

1. patient who refuses oophorectomy
2. medical condition in which surgery cannot be tolerated Any waiver of these inclusion and exclusion criteria must be approved by the investigator on a case-by case basis prior to enrolling the subject. This must be documented by the investigator. No subject will be allowed to enroll in this study more than once.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Disease free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Won-Suk Lee, M.D., Principal Investigator — Gachon Univ. GIl Hospital
Locations (1):
- Won-Suk Lee, Incheon, Incheon, South Korea

REFERENCES:
- [Background] Moore RG, Chung M, Granai CO, Gajewski W, Steinhoff MM. Incidence of metastasis to the ovaries from nongenital tract primary tumors. Gynecol Oncol. 2004 Apr;93(1):87-91. doi: 10.1016/j.ygyno.2003.12.039. PMID 15047218